CLINICAL TRIAL: NCT04378270
Title: Validation of a Novel Foot Offloading Device
Acronym: PopSole2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey A. Gusenoff, MD (Other)
Responsible Party: Sponsor-Investigator, Jeffrey A. Gusenoff, MD, Professor of Plastic Surgery, & Director, Foot Fat Grafting Institute, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20010059
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fasciitis, Chronic; Heel Pain Syndrome; Fat Pad Syndrome
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PopSole™ offloading device (Experimental): This is an external insole device that fits into a shoe and is reusable for a given subject, not for one-time use. It is comparable to other off-the-shelf insoles readily available and presents minimal risk to the participant during the four weeks of study participation.
  Interventions: Device: PopSole™ Offloading Device

INTERVENTIONS:
Device: PopSole™ Offloading Device — Specifically, the PopSole™ Offloading Device allows the provider to pop bubbles in the device (like popping paper or plastic bubble sheeting), thereby offloading the surgical area or area of pain. This customizable approach to offloading may increase compliance as it can easily fit in a normal walking shoe and is personalized for each patient. It can also be attached to a slide for use in the shower. Currently no post-operative devices for offloading the foot can be used in the shower.

SUMMARY:
Pressure offloading is often considered the most crucial aspect in healing after a foot injury. The investigators have devised a novel foot offloading device (PopSole™) which will allow for customization of the area where there is foot pain, as well as allow for customizable arch support and elevation of the metatarsals. This validation study is aimed to assess improvement of pain with use, ease of use, fit and feel, compliance, and durability over a 4 week period. Validated patient reported outcome measures will be used at baseline, 2 weeks and 4 weeks.

DETAILED DESCRIPTION:
All subjects will receive the PopSole™ offloading device at the screening/baseline visit, be asked to wear it for 4 weeks, and will be asked to return for an in-person evaluation at week 2 and a completion study visit at week 4.

Screening includes the following procedures:

1. Performance of a limited physical exam, inclusive of participant's foot exam with a gait and shoe gear evaluation.
2. Medical and surgical history collection
3. Vital signs, medication profile, allergies, height, weight, and BMI calculation.
4. Collection of demographic information
5. 2D Photographs of both feet will be performed

Subjects will be asked to complete:

1. Questionnaires

   * Foot and Ankle Ability Measure questionnaire
   * Mayo Clinical Scoring System questionnaire
   * American Orthopaedic Foot and Ankle Society questionnaire
   * Manchester Foot and Ankle Disability Index
   * Pittsburgh Foot Survey
2. Diary cards to document for the feet: pain, bruising, redness of the skin, itching, swelling, bleeding, and any concerns/issues not listed, as well as the location, date and day for each noted symptom.
3. Offload Device Distribution. Devices will be provided for both feet to maintain symmetry and gait stability between the two feet. One pair of devices will be given for use in shoe gear, and one pair will be given for use in a slide in the shower.

Follow up visit procedures:

Week 2

1. Collection of vital signs, medication profile, weight, and BMI calculation
2. Limited physical exam with a foot exam
3. Adverse Event Reporting
4. Collection and distribution of feet diary cards
5. 2D Photographs of both feet
6. Foot Assessment Questionnaires
7. Device survey - questions about the fit and feel of the device

Week 4

The same procedures listed for week 2, with the addition of PopSole™ Device removal and final foot diary card collection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Subjects with foot pain due to forefoot or heel fat pad atrophy or chronic plantar fasciitis as defined by heel pain for greater than 6 months and failed non-surgical therapy
3. Willing and able to comply with follow up examinations

Exclusion Criteria:

1. Concurrent injury to the lower extremity that would effect gait
2. Open foot ulcerations, fractures, or diagnosis of osteomyelitis of the feet
3. Surgical foot intervention in the last 6 months
4. Diagnosis of pregnancy or the intent of the participant to become pregnant during participation in this study
5. Neuropathy
6. Any issue that per the physician's determination would render the patient not appropriate to continue participation in the study (compliance, change in physical status, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gusenoff, MD, Principal Investigator — Professor of Plastic Surgery, Director of the Foot Fat Grafting Institute
Locations (1):
- UPMC Aesthetic Plastic Surgery Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gusenoff JA, Mitchell RT, Jeong K, Wukich DK, Gusenoff BR. Autologous Fat Grafting for Pedal Fat Pad Atrophy: A Prospective Randomized Clinical Trial. Plast Reconstr Surg. 2016 Nov;138(5):1099-1108. doi: 10.1097/PRS.0000000000002667. PMID 27391833
- [Background] Minteer DM, Gusenoff BR, Gusenoff JA. Fat Grafting for Pedal Fat Pad Atrophy in a 2-Year, Prospective, Randomized, Crossover, Single-Center Clinical Trial. Plast Reconstr Surg. 2018 Dec;142(6):862e-871e. doi: 10.1097/PRS.0000000000005006. PMID 30204683
- [Background] Swinnen E, Kerckhofs E. Compliance of patients wearing an orthotic device or orthopedic shoes: A systematic review. J Bodyw Mov Ther. 2015 Oct;19(4):759-70. doi: 10.1016/j.jbmt.2015.06.008. Epub 2015 Jul 2. PMID 26592234
- [Background] Jarl G. Methodological considerations of investigating adherence to using offloading devices among people with diabetes. Patient Prefer Adherence. 2018 Sep 12;12:1767-1775. doi: 10.2147/PPA.S175738. eCollection 2018. PMID 30254428
- [Background] Waaijman R, Keukenkamp R, de Haart M, Polomski WP, Nollet F, Bus SA. Adherence to wearing prescription custom-made footwear in patients with diabetes at high risk for plantar foot ulceration. Diabetes Care. 2013 Jun;36(6):1613-8. doi: 10.2337/dc12-1330. Epub 2013 Jan 15. PMID 23321218
- [Background] Polat G, Karademir G, Akalan E, Asik M, Erdil M. Patient compliance with touchdown weight bearing after microfracture treatment of talar osteochondral lesions. J Orthop Surg Res. 2017 Mar 20;12(1):46. doi: 10.1186/s13018-017-0548-5. PMID 28320425
- [Background] Arts ML, de Haart M, Bus SA, Bakker JP, Hacking HG, Nollet F. Perceived usability and use of custom-made footwear in diabetic patients at high risk for foot ulceration. J Rehabil Med. 2014 Apr;46(4):357-62. doi: 10.2340/16501977-1272. PMID 24356801
- [Background] Bus SA, van Deursen RW, Kanade RV, Wissink M, Manning EA, van Baal JG, Harding KG. Plantar pressure relief in the diabetic foot using forefoot offloading shoes. Gait Posture. 2009 Jun;29(4):618-22. doi: 10.1016/j.gaitpost.2009.01.003. Epub 2009 Feb 13. PMID 19217785
- [Background] Wunnemann M, Klein D, Rosenbaum D. Effects of the Twin Shoe (Darco) to compensate height differences in normal gait. Gait Posture. 2011 Jan;33(1):61-5. doi: 10.1016/j.gaitpost.2010.09.025. Epub 2010 Oct 20. PMID 20961763
- [Background] Myers KA, Long JT, Klein JP, Wertsch JJ, Janisse D, Harris GF. Biomechanical implications of the negative heel rocker sole shoe: gait kinematics and kinetics. Gait Posture. 2006 Nov;24(3):323-30. doi: 10.1016/j.gaitpost.2005.10.006. Epub 2005 Nov 21. PMID 16300949
- [Background] Braun BJ, Veith NT, Rollmann M, Orth M, Fritz T, Herath SC, Holstein JH, Pohlemann T. Weight-bearing recommendations after operative fracture treatment-fact or fiction? Gait results with and feasibility of a dynamic, continuous pedobarography insole. Int Orthop. 2017 Aug;41(8):1507-1512. doi: 10.1007/s00264-017-3481-7. Epub 2017 Apr 19. PMID 28421239
- [Background] Bus SA, Maas JC, Otterman NM. Lower-extremity dynamics of walking in neuropathic diabetic patients who wear a forefoot-offloading shoe. Clin Biomech (Bristol). 2017 Dec;50:21-26. doi: 10.1016/j.clinbiomech.2017.10.003. Epub 2017 Oct 2. PMID 28985487
- [Background] Robinson C, Major MJ, Kuffel C, Hines K, Cole P. Orthotic management of the neuropathic foot: an interdisciplinary care perspective. Prosthet Orthot Int. 2015 Feb;39(1):73-81. doi: 10.1177/0309364614545422. PMID 25614503
- [Background] Jarl G, Tranberg R. An innovative sealed shoe to off-load and heal diabetic forefoot ulcers - a feasibility study. Diabet Foot Ankle. 2017 Jul 25;8(1):1348178. doi: 10.1080/2000625X.2017.1348178. eCollection 2017. PMID 28804593
- [Background] de Oliveira AL, Moore Z. Treatment of the diabetic foot by offloading: a systematic review. J Wound Care. 2015 Dec;24(12):560, 562-70. doi: 10.12968/jowc.2015.24.12.560. PMID 26654736
- [Background] Bus SA. The Role of Pressure Offloading on Diabetic Foot Ulcer Healing and Prevention of Recurrence. Plast Reconstr Surg. 2016 Sep;138(3 Suppl):179S-187S. doi: 10.1097/PRS.0000000000002686. PMID 27556758
- [Background] Janisse DJ, Janisse E. Shoe modification and the use of orthoses in the treatment of foot and ankle pathology. J Am Acad Orthop Surg. 2008 Mar;16(3):152-8. doi: 10.5435/00124635-200803000-00006. PMID 18316713
- [Background] Farber SE, Minteer D, Gusenoff BR, Gusenoff JA. The Influence of Fat Grafting on Skin Quality in Cosmetic Foot Grafting: A Randomized, Cross-Over Clinical Trial. Aesthet Surg J. 2019 Mar 14;39(4):405-412. doi: 10.1093/asj/sjy168. PMID 30007274
- [Result] Lubarsky R, Gusenoff B, Gusenoff JA. Prospective Cohort Validation Study of a Novel Foot Offloading Device. Plast Reconstr Surg Glob Open. 2021 Nov 24;9(11):e3950. doi: 10.1097/GOX.0000000000003950. eCollection 2021 Nov. PMID 34840921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants were recruited to a 1 month cohort, and 10 participants to a 3 month cohort.
Pre-assignment Details: 1 participant was a screen failure and was not found eligible to continue to intervention.
Period: Overall Study
Arm/Group | PopSole™ Offloading Device
Started | 20
Completed | 15
Not Completed | 5
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Screen Failure | 1
Not completed — University Required, Research Covid Shut Down | 2

BASELINE CHARACTERISTICS:
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Number of participants who received PopSole device at baseline [Count of Participants; unit: Participants] | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Foot Pain From Screening/Baseline Visit to 4 Week Visit as Reported on the Pittsburgh Foot Survey.
Description: Pain and function questionnaire measure. Scale for pain ranges from "Very severe" to "Had no pain". Scale for pain interference ranges from " Very much" to "not at all". Scale of functionality ranges from "unable to do" to "without any difficulty" in regards to a range of specified activities. Change is reported in mean foot reported pain score Screening/Baseline visit to 4 Week visit. Questions related to pain include items 1-5, total pain score possible is 25; higher scores indicate less pain reported.
Time Frame: Four Weeks
Population: 19 participants received the study device, 15 completed a 4 week visit.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 15
Score on a scale | 2.930 [-0.3687 to 6.2287]
Statistical Analysis 1: Comparison: PopSole™ Offloading Device; This procedure calculates the difference between the observed means in two independent samples (two collected assessment timepoints, screening and 4 week follow up visits). A significance value (P-value) and 95% Confidence Interval (CI) of the difference is reported. The P-value is the probability of obtaining the observed difference between the samples if the null hypothesis were true. The null hypothesis is the hypothesis that the difference is 0; Test type: Other; p = 0.0796, t-test, 2 sided; Degrees of Freedom (DF)- 28; Mean Difference (Final Values) = 2.930, 95% CI 2-sided [-0.3687 to 6.2287], Standard Error of Mean 1.610

2. Primary Outcome: Change in Foot Pain From Screening/Baseline Visit to 4 Week Visit as Reported on the Manchester Foot and Ankle Index.
Description: Pain and function questionnaire assessment. Three responses to a variety of pain and specified activities raging from "On most/every day(s)" which is scored as 2 to "none of the time" which is scored as 0. Summation is made on Functional (0-20 with 20 being the lowest functioning), Personal appearance (0-4 with 4 being the worst), pain (0-10 with 10 being the worst), work/leisure (0-100 with 100 being the worst impact on work/leisure).
  Change in mean foot pain as reported on the Manchester Foot and Ankle Index from Screening/Baseline visit to 4 Week visit. Pain subscale is questions 13-17, range is 0-10 total points, lower scores indicate less pain.
Time Frame: Four Weeks
Population: 19 participants received the study device, 15 completed a 4 week visit.
Measure: Mean (95% Confidence Interval); unit: Score on a scale.
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 15
Score on a scale. | -1.7 [-3.5014 to 0.1014]
Statistical Analysis 1: Comparison: PopSole™ Offloading Device; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0634, t-test, 2 sided; Degrees of Freedom (DF)- 28; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.5014 to 0.1014], Standard Error of Mean 0.879

3. Primary Outcome: Change in Foot Pain From Screening/Baseline Visit to 4 Week Visit as Reported on the Mayo Clinical Scoring System Questionnaire.
Description: Pain and function questionnaire. Pain scale from 0 (worst) to 50 (no pain). Activity limitations, orthotic requirements, antalgic gait, neuropathy and plantar heel tenderness are all graded 10 (best) to 10 (worst). Overall summation is excellent (90-100), good (80-89), fair (70-79), poor (<70).
  Change in mean foot pain score on Mayo Clinical Scoring System Questionnaire from Screening/Baseline Visit to 4 Week Visit. Pain scale is the first question, 50 total points, with higher scores meaning less pain.
Time Frame: Four Weeks
Population: 19 participants received the study device. 15 completed a 4 Week visit.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 15
score on a scale | 18.7 [7.4498 to 29.9502]
Statistical Analysis 1: Comparison: PopSole™ Offloading Device; This procedure calculates the difference between the observed means in two independent samples (two collected assessment timepoints, screening and 4 week follow up visits). A significance value (P-value) and 95% confidence interval (CI) of the difference is reported. The P value is the probability of obtaining the observed difference between the samples if the null hypothesis were true. The null hypothesis is the hypothesis that the difference is 0; Test type: Other; p = 0.0020, t-test, 2 sided; Degrees of Freedom (DF)- 28; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [7.4498 to 29.9502], Standard Error of Mean 5.492

4. Primary Outcome: Change in Foot Pain From Screening/Baseline Visit to 4 Week Visit as Reported on the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale.
Description: This survey assesses pain (40 points possible, comprises pain subtotal), function (50 points possible, comprises function subtotal; which includes activity limitations, maximum walking distance, difficulty with walking surfaces, gait abnormality, sagittal motion, hindfoot motion and ankle/hindfoot stability, and alignment (10 possible points, comprises alignment subtotal). A total score is calculated out of 100, with higher scores indicating greater impairment. There are also calculated subtotals specific to pain, function and alignment.
  Change in mean foot pain score on AOFAS from Screening/Baseline Visit to 4 Week Visit. Pain scale is 40 total points, with higher scores meaning less pain.
Time Frame: Four Weeks
Population: 19 participants received the study device. 15 completed a 4 Week visit.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 15
score on a scale | 16.67 [7.8069 to 25.5331]
Statistical Analysis 1: Comparison: PopSole™ Offloading Device; Test type: Other; p = 0.0006, t-test, 2 sided; Degrees of freedom (DF)- 28; Mean Difference (Net) = 16.67, 95% CI 2-sided [7.8069 to 25.5331], Standard Error of Mean 4.327

5. Primary Outcome: Device Durability
Description: Documentation of the number of participants who wore a single device for first 4 weeks of the participant's study participation.
Time Frame: Four weeks.
Population: 19 participants received the study device at baseline. 1 participant withdrew prior to the four week, 2 participants were withdrawn from the study due to the University of Pittsburgh's ordered research shutdown due to Covid, and one participant missed the four week visit.
Measure: Count of Participants; unit: Participants
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 19
Participants | 15

6. Primary Outcome: Participant Compliance With Device
Description: Documentation of the number of participants who did not wear a single device for the full 4 weeks of the participant's study participation.
Time Frame: Four Weeks
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 19
Participants | 4

7. Secondary Outcome: Participants' Reported Satisfaction and/or Difficulties With the Device
Description: As measured by subject self report, using a device satisfaction measure questionnaire. Questions are answered yes/no in all cases except comfort (1-10 with 10 being the most comfortable), and ease of use (1-10 with 10 being most easy to use).
Time Frame: Four Weeks
Population: Participants reported comfort with the PopSole Device on a 1-10 scale, 1= very uncomfortable and 10=very comfortable. Participants reported on the ease of using the PopSole Device on 1-10 scale, 1=very difficult and 10=very easy. 20 total points possible, higher score indicates increased satisfaction.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PopSole™ Offloading Device
Number analyzed (Participants) | 15
score on a scale | 17.87 (2.39)
Statistical Analysis 1: Comparison: PopSole™ Offloading Device; This procedure calculates the difference of an observed mean (from the assessment collected at the 4 week visit) with a hypothesized mean value (10, a mid level scale score). A significance value (P-value) and 95% Confidence Interval (CI) of the observed mean is reported. The P-value is the probability of obtaining the observed mean in the sample if the null hypothesis value were the true value; Test type: Other; p = 0.0001, t-test, 2 sided; Degrees of freedom (DF)- 14; Mean pain scale = 17.87, 95% CI 2-sided [16.5465 to 19.1935], Standard Deviation 2.39

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each timepoint, over a period of 1 month for the first cohort, and over a period of 3 months for the second cohort.
Arm/Group | PopSole™ Offloading Device
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PopSole™ Offloading Device (N=20)
pain at left metatarsal on left foot (General disorders) | 1 (1) — Subject reported moderate pain to investigators, determined to be unrelated to Popsole device, resolved without sequelae within 2 days of onset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04378270/Prot_SAP_001.pdf